CLINICAL TRIAL: NCT04696172
Title: Explore Potential Plasma Biomarkers of Acute Respiratory Distress Syndrome (ARDS) Using Proteomics Analysis in Patients Undergoing Cardiopulmonary Bypass
Brief Title: Plasma Biomarkers of Cardiopulmonary Bypass Induced Acute Respiratory Distress Syndrome (CPB-ARDS)
Acronym: PBOARDS
Status: Completed | Type: Observational
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Wuhan Asia Heart Hospital (Other)
Responsible Party: Principal Investigator, Shanglong Yao, Clinical Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: V1.0
Record Dates: First submitted 2020-12-28; First posted 2021-01-06 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Acute Respiratory Distress Syndrome; Biomarkers; Proteomics; Cardiopulmonary Bypass
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Biospecimen Retention: Samples With DNA — Plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients undergoing cardiopulmonary bypass (CPB) with postoperative ARDS
- Patients undergoing cardiopulmonary bypass (CPB) without postoperative ARDS

SUMMARY:
The investigators aimed to establish a prospective cohort of patients undergoing cardiopulmonary bypass (CPB) in cardiac surgery from April 2021 to September 2022, in Wuhan. The ARDS events, ventilation time, time of extubation, oxygenation index for 3 days after operation were observed. Plasma samples were collected before CPB, and several time points after CPB. Dynamic differential proteins of ARDS after CPB were screened by DIA (Data independent acquisition) proteomics. Quantitative protein marker concentration was used to predict the occurrence of ARDS after operation, the model discrimination and calibration was assessed.

ELIGIBILITY:
Inclusion Criteria:

* Selective operation;
* Cardiac surgery with cardiopulmonary bypass;
* Adult patients over 18 years old;
* Signed informed consent

Exclusion Criteria:

* patients who refuse to sign the informed consent form or the attending physician refuses the patient to join the study;
* non elective surgery (surgery at non-elective time or emergency surgery);
* preoperative pulmonary insufficiency, pulmonary hypertension and pulmonary inflammation;
* the absence of any specimen and clinical data;
* patients who failed the operation, needed extracorporeal membrane oxygenation support or underwent CPB operation again within 3 days after operation;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiopulmonary bypass (CPB) in cardiac surgery from April 2021 to July 2022, in Wuhan Union hospital
Sampling Method: Probability Sample
Enrollment: 525 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with postoperative ARDS events as assessed by Berlin Definition. | 3 days after operation
  The Berlin Definition of Acute Respiratory Distress Syndrome:
  1. Timing: Within 1 week of a known clinical insult or new or worsening respiratory symptoms;
  2. Chest imaging: Bilateral opacities-not fully explained by effusions, lobar/lung collapse, or nodules;
  3. Origin of edema: Respiratory failure not fully explained by cardiac failure or fluid overload. Need objective assessment (eg, echocardiography) to exclude hydrostatic edema if no risk factor present;
  4. Oxygenation:
  Mild 200 mm Hg <PaO2/FIO2≤ 300 mm Hg with PEEP or CPAP ≥5 cm H2O; Moderate 100 mm Hg <PaO2/FIO2≤ 200 mm Hg with PEEP ≥5 cm H2O Severe PaO2/FIO2≤ 100 mm Hg with PEEP ≥5 cm H2O

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Wuhan Asia Heart Hospital, Wuhan, Hubei

REFERENCES:
- [Derived] Wang Y, Chen L, Yao C, Wang T, Wu J, Shang Y, Li B, Xia H, Huang S, Wang F, Wen S, Huang S, Lin Y, Dong N, Yao S. Early plasma proteomic biomarkers and prediction model of acute respiratory distress syndrome after cardiopulmonary bypass: a prospective nested cohort study. Int J Surg. 2023 Sep 1;109(9):2561-2573. doi: 10.1097/JS9.0000000000000434. PMID 37528797